CLINICAL TRIAL: NCT02916043
Title: Risk Factor of Acute Kidney Injury After Open Heart Surgery With Cardiopulmonary Bypass
Brief Title: Neutrophil, Lymphocyte and Platelet as a Predictor for AKI and Mortality
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Won Ho Kim, MD, Clinical Associate Professor, Seoul National University Hospital
Other Study IDs: 1604-038-753
Record Dates: First submitted 2016-09-25; First posted 2016-09-27 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-09

CONDITIONS: Acute Kidney Injury
Keywords: acute kidney injury; cardiovascular surgery; mortality
MeSH Terms: conditions — Acute Kidney Injury | interventions — Cardiovascular Surgical Procedures; Cardiopulmonary Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Cardiovascular surgery with cardiopulmonary bypass: Cardiovascular surgery with cardiopulmonary bypass
  Interventions: Procedure: Cardiovascular surgery with cardiopulmonary bypass

INTERVENTIONS:
Procedure: Cardiovascular surgery with cardiopulmonary bypass — Patients who underwent cardiovascular surgery including valve replacement or thoracic aortic surgery with cardiopulmonary bypass

SUMMARY:
Cell-count related risk factors for acute kidney injury after cardiovascular surgery have been reported. The authors attempted to investigate whether the perioperative cell counts of neutrophil, lymphocyte, platelet are associated with the postoperative acute kidney injury and long-term mortality after cardiovascular surgery using cardiopulmonary bypass.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) after cardiovascular surgery remains a serious complication associated with increased mortality for up to 10 years. The incidence of AKI after cardiovascular surgery is as high as 55% and the incidence of renal replacement therapy (RRT) to be up to 8 %.

Cell-count related risk factors for acute kidney injury after cardiovascular surgery have been reported. The authors attempted to investigate whether the perioperative cell counts of neutrophil, lymphocyte, platelet are associated with the postoperative acute kidney injury and long-term mortality after cardiovascular surgery using cardiopulmonary bypass.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who underwent cardiovascular surgeries with cardiopulmonary bypass (CPB), including valve replacement and surgery on the thoracic aorta at the Seoul National University Hospital between 2007 and 2015

Exclusion Criteria:

* Missing preoperative serum creatinine (sCr) values
* Missing preoperative platelet, neutrophil and lymphocyte counts
* Patients who underwent preoperative hemodialysis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients who underwent cardiovascular surgeries with cardiopulmonary bypass (CPB), including valve replacement and surgery on the thoracic aorta at the Seoul National University Hospital between 2007 and 2015
Sampling Method: Non-Probability Sample
Enrollment: 1099 (Actual)
Dates: Start 2016-04; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Acute kidney injury | postoperative day seven
  acute kidney injury during postoperative seven days defined by Kidney Disease Improving Global Outcomes (KDIGO) criteria

SECONDARY OUTCOMES:
All-cause mortality | postoperative seven years
  all-cause mortality after cardiovascular surgery after postoperative seven years

OTHER OUTCOMES:
Postoperative length of hospital stay | postoperative two month
  postoperative length of hospital stay
Postoperative length of ICU stay | postoperative two months
  postoperative length of ICU stay during postoperative two months
Postoperative incidence of complications | postoperative two months
  postoperative incidences of surgery-related complications during hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No